CLINICAL TRIAL: NCT07149311
Title: Effectiveness of Diabetes Self-management Education on Diabetes Control in Patients With Type 2 Diabetes Mellitus: A Randomized Controlled Trial
Brief Title: Effectiveness of Diabetes Self-management Education on Glycaemic Control in Patients With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Komfo Anokye Teaching Hospital (Other)
Responsible Party: Principal Investigator, Kojo Awotwi Hutton-Mensah, Doctor, Komfo Anokye Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KATHIRB/AP/106/23
Record Dates: First submitted 2025-07-02; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Diabete Type 2
Keywords: diabetes self management education; effectiveness; glycaemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group that received only usual care (Control ) (No Intervention): The current standard practice (the usual care) includes an outpatient specialist service with patients scheduled every 1 to 6 months, depending on their diabetes control and complications profile. The other services provided include dietician appointments, laboratory investigations, clinical examinations, group education on self-management practices, and medication refills.
  Usual care by a doctor entails a 10-15 min standard doctors' consultation where the recent HbA1c level and medication compliance are reviewed, and a brief informal patient-tailored diabetes education is offered. This enables the individual an opportunity to learn about self-management in a flexible and informal way. There is no structure to it and the information is offered according to what the patient requests to know as well as what the doctor thinks would be important for the patient to know, during that consultation.
  Phone calls will be made to remind them of their clinic appointment for data collection.
- Group that received DSME plus usual care (Intervention) (Experimental): The intervention group will receive the usual consultation from their doctor and referral to a diabetes educator for individualized structured DSME training. A clinical sheet will be used while delivering the education to ensure that all core topics are covered. For this study, 2 diabetes educators will offer the individualized DSME sessions using the American Association of Diabetes Education (AADE) 7 self-care behaviour model. The participants are scheduled to attend a 1-hour individualised session at the hospital every 3 months as well as telephone consultations lasting up to 15 minutes every 2 weeks at the convenience of the participant to reinforce DSME for 6 months. The first session is arranged on the first day after consultation with the doctor. At the end of the sessions, the participants will receive a patient guide to diabetes booklet and graphic material illustrating several self-care activities such as foot care
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — The intervention group will receive the usual consultation from their doctor and referral to a diabetes educator for individualised structured DSME training. A clinical sheet will be used while delivering the education to ensure that all core topics are covered. For this study, 2 diabetes educators will offer the individualised DSME sessions using the American Association of Diabetes Education (AADE) 7 self-care behaviour model. The participants are scheduled to attend a 1-hour individualised session at the hospital every 3 months as well as telephone consultations lasting up to 15 minutes every 2 weeks at the convenience of the participant to reinforce DSME for 6 months. The first session is arranged on the first day after consultation with the doctor. At the end of the sessions, the participants will receive a patient guide to diabetes booklet and graphic material illustrating several self-care activities such as foot care
  Arms: Group that received DSME plus usual care (Intervention)

SUMMARY:
This is a randomized controlled trial assessing the effectiveness of a nurse led diabetes self management education(DSME) given over a 6 month period via mixed delivery strategy (in-person and via phone calls) on Hemoglobin A1c(HbA1c), fasting blood glucose(FBG), blood pressure, body weight and low density lipoprotein cholesterol(LDL-C).

The main question this research seeks to answer is

1. Does diabetes self-management education when combined with usual care improve glycaemic control when compared to usual care alone? Patients will be randomized into intervention and control groups. The intervention group will receive nurse led DSME using the American Association of diabetes educators 7 self care behaviour over a 6 month period. It will involve 3 monthly in-person sessions starting from the first day of recruitment as well as 2 weekly phone call sessions. This will be in addition to the usual care at the diabetes clinic.

The control group will receive usual diabetes care

DETAILED DESCRIPTION:
This a randomized controlled parallel design among 74 Type 2 diabetes mellitus(T2DM) patients recruited from the Komfo Anokye Teaching Hospital Diabetes clinic.

The primary outcome is the mean change in HbA1c at 6 months

The secondary outcomes include:

1. The mean change in FBG at 3 months
2. The mean change in blood pressure at 6 months
3. The mean change in body weight at 6 months
4. The mean change in LDL-C at 6 month

STUDY PROTOCOL USUAL CARE The current standard practice (the usual care) includes an outpatient specialist service with patients scheduled every 1 to 6 months, depending on their diabetes control and complications profile. The other services provided include dietician appointments, laboratory investigations, clinical examinations, group education on self-management practices, and medication refills.

Usual care by a doctor entails a 10-15 min standard doctors' consultation where the recent HbA1c level and medication compliance are reviewed, and a brief informal patient-tailored diabetes education is offered. This enables the individual an opportunity to learn about self-management in a flexible and informal way. There is no structure to it and the information is offered according to what the patient requests to know as well as what the doctor thinks would be important for the patient to know, during that consultation.

Phone calls will be made to remind them of their clinic appointment for data collection.

THE INTERVENTION- DIABETES SELF-MANAGEMENT EDUCATION The intervention group will receive the usual consultation from their doctor and referral to a diabetes educator for individualized structured DSME training. An empowerment and interactive teaching model will be used with focus on behavioral assessment, goal-setting and problem-solving to promote autonomous self-regulation for better health and quality of life. A clinical sheet will be used while delivering the education to ensure that all core topics are covered.

For this study, 2 diabetes educators will offer the individualized DSME sessions using the American Association of Diabetes Education (AADE) 7 self-care behaviour model which focuses on: being active, healthy eating, monitoring blood glucose, healthy coping, reducing risks, problem solving and adherence to medication The participants are scheduled to attend a 1-hour individualized session at the hospital every 3 months as well as telephone consultations lasting up to 15 minutes every 2 weeks at the convenience of the participant to reinforce DSME for 6 months. The first session is arranged on the first day after consultation with the doctor. At the end of the sessions, the participants will receive a patient guide to diabetes booklet and graphic material illustrating several self-care activities such as foot care . Subsequent consultations will be mainly feedback sessions, aimed at reviewing previously discussed matters, reinforcing key messages, addressing challenges and providing additional information.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM who are at least 18 years old without any co-morbidities requiring immediate hospitalisation
* HbA1c >7.9%
* Have access to a personal mobile phone and able to answer calls.
* Mentally stable, with no vision, verbal, or hearing impairments
* Have access a glucometer.
* Consents to the study

Exclusion Criteria:

* Other forms of DM such as type 1 DM or gestational diabetes.
* End-stage renal disease(eGFR<15ml/min)
* Anaemia
* History of stroke or other atherosclerotic cardiovascular diseases with impairment which makes the affected individual dependent on others for care giving and precludes self-care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Primary outcome measuring the mean change in HbA1c at 6 months | 6 months
  Mean change in HbA1c

SECONDARY OUTCOMES:
Secondary outcome measuring the mean change in fasting blood glucose at 3 months | 3 months
  Mean change in fasting blood glucose 2) The mean change in blood pressure at 6 months 3) The mean change in body weight at 6 months 4) The mean change in LDL-C at 6 month
Secondary outcome measuring the mean change in blood pressure at 6 months | 6 months
  Mean change in blood pressure
Secondary outcome measuring the mean change in body weight at 6 months | 6 months
  Mean change in body weight
Secondary outcome measuring the mean change in low density lipoprotein cholesterol at 6 months | 6 months
  Mean change in low density lipoprotein cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- Komfo Anokye Teaching Hospital, Kumasi, Ghana

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT07149311/Prot_SAP_000.pdf